CLINICAL TRIAL: NCT06650267
Title: Substance Misuse and Family Violence Treatment for Fathers
Brief Title: Substance Misuse and Family Violence Treatment Fathers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: APT Foundation, Inc. (Other); VA Connecticut Healthcare System (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000038147; 1R01DA059914-01A1 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Substance Misuse; Violence, Domestic; Child Abuse
Keywords: substance misuse; intimate partner violence; domestic violence; treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fathers for Change (Experimental)
  Interventions: Behavioral: Fathers for Change (F4C)
- Individual Drug Counseling (Active Comparator)
  Interventions: Behavioral: Individual Drug Counseling (IDC)

INTERVENTIONS:
Behavioral: Fathers for Change (F4C) — Defining features of F4C delivered over 18 sessions: 1) focus on the fathers model of fatherhood as a motivator for change, 2) focus on understanding and identifying feelings, teaching skills to identify and change emotional dysregulation that lead to both SU and FV, 3) co-parent communication skills to reduce stress and improve problem solving, 4) restorative parenting (see Table 1 and figure 1)127. F4C focuses on reflective understanding of emotional experiences, how that impacts thoughts and behaviors related to SU, FV, co-parenting/parenting each session. Through greater self-awareness, the father is better able to apply coping, communication and parenting skills introduced to reduce SU and FV.
  Arms: Fathers for Change
Behavioral: Individual Drug Counseling (IDC) — IDC is an individual evidence-based SU treatment84 that incorporates two elements: endorsement of the disease model and the spiritual dimensions of recovery. These elements differentiate the approach from F4C. IDC is influenced by 12-step recovery philosophy and participation in 12-step groups like NA are encouraged. The model places focus on the individual in recovery without a focus on fatherhood or co-parenting. IDC will be offered in an 18-session format.
  Arms: Individual Drug Counseling

SUMMARY:
This study involves a randomized controlled trial of Fathers for Change (F4C) compared to Individual Drug Counseling (IDC) with a sample of 280 fathers enrolled in substance use (SU) treatment within community or veterans (VA) healthcare settings to (a) demonstrate F4C efficacy compared to IDC in reducing SU and family violence (FV) at end of treatment, 3- and 6-month post-treatment follow-up, and (b) document improved emotion regulation as the mechanism within F4C that results in reduced SU and FV.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM-5 criteria for an SU disorder at the time of assessment at APT or VACHS;
* report FV within the last 18 months prior to screening (based on self, court, police or child protection reports);
* have at least one biological child aged 1 to 12 years with whom they live or have at least twice per month in person visits;
* are able to complete assessments in English; and
* agree to have their female coparents (mother of the youngest child) contacted for participation of their youngest child. If a participant has more than one child in the age range, the youngest will be the target of assessment and treatment.

Exclusion Criteria:

* an active full/no contact protective order pertaining to their child;
* physiological addiction to a substance that requires detoxification (such individuals may be re-evaluated following detox);
* cognitive impairment (a mini mental state score <25);
* current untreated psychotic/bipolar disorder;
* currently suicidal or homicidal based on Brief Symptom Inventory Screening and follow-up on positive responses; or
* are currently receiving weekly individual therapy for Substance misuse or family violence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Substance Misuse | Baseline (week 0), weekly during treatment for through 18 week, Post-Treatment at week 19, week 32 and week 45
  Self-reported days of substance misuse reported a positive breathalyzer/urine tox screen will be used to create a sum of the number of weeks with use during treatment and at each follow-up period.
Family Violence (FV) | Baseline (week 0), weekly during treatment for through 18 week, Post-Treatment at week 19, week 32 and week 45
  Any instance of FV either toward a partner or child identified by any report (self-report on the Timeline Followback weekly surveys, child protection or arrest record) will be counted to allow for the best estimate of FV across reports resulting in a sum count of the number of FV incidents during the 18 weeks of treatment and from post-treatment to each follow-up timepoint

SECONDARY OUTCOMES:
Emotion Dysregulation | Baseline (week 0), Post-Treatment at week 19, week 32 and week 45
  The Difficulties in Emotion Regulation Scale will be used to measure self-reported emotion regulation. Sum scores range from 18 to 90 with higher scores suggesting more impaired emotion regulation.
Articulated Thoughts in Simulated Situations (ATSS) | Baseline (week 0) and Post-Treatment (week 18)
  The participants responses to the ATSS will be coded for hostile responding and will serve as a non-self-report measure of emotion regulation. Scores range from 0 to 5 with 5 being greater hostile responding across scenarios.

CONTACTS AND LOCATIONS:
Overall Officials: Carla S Stover, Ph.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University Child Study Center, New Haven, Connecticut
  - APT Foundation, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Clinical/assessment data will be deposited into Harvard Dataverse at the conclusion of study data collection and publication of primary study specific aims.
Supporting Information: Study Protocol
Time Frame: The research community will have access to data when the primary analyses have been completed and published.
Access Criteria: Researchers will request access to the data through a standard request and approval by the study PI and then release by the repository